CLINICAL TRIAL: NCT00330928
Title: Coronary Artery Plaque Characterization by NIR Spectroscopy in Patients Undergoing Elective Percutaneous Coronary Intervention
Brief Title: SPECTACL: SPECTroscopic Assessment of Coronary Lipid
Acronym: SPECTACL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Infraredx (Industry)
Responsible Party: Director of Clinical & Regulatory Affairs, InfraReDx Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0101; CL0101
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Results first posted 2009-05-28 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Angina Pectoris; Angina, Unstable; Myocardial Infarction
MeSH Terms: conditions — Angina Pectoris; Angina, Unstable; Myocardial Infarction | interventions — Spectroscopy, Near-Infrared; Diagnostic Imaging; Ultrasonography, Interventional

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Subjects undergoing elective percutaneous coronary intervention
  Interventions: Device: Near Infrared Spectroscopy (NIRS) Imaging; Device: intravascular ultrasound (IVUS)

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) Imaging — Near infrared spectroscopic imaging of the coronary artery with an intravascular spectroscopy catheter.
  Other Names: InfraReDx, LipiScan (prototype)
Device: intravascular ultrasound (IVUS) — Ultrasound coronary catheter is positioned on a guidewire that has been placed in the coronary artery.Ultrasound imaging provides structural information about the vessel wall and blockages contained. It takes approximately 5 minutes to prepare, position, and to collect data with the catheter.
  Other Names: Volcano, Revolution; Volcano, Eagle Eye; Boston Scientific, Atlantis

SUMMARY:
The purpose of this study is to evaluate a near-infrared (NIR) spectroscopy system that has been designed to identify the chemical composition of coronary artery plaques in patients undergoing a percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Extensive studies conducted over the past 7 years in autopsy specimens have demonstrated that NIR spectroscopy can identify the plaque structures that are suspected to cause the acute coronary artery syndromes(unstable angina, myocardial infarction, and sudden death).

The application of NIR spectroscopy to identify lipid deposition within coronary arteries has shown promising results in preclinical ex vivo studies (14). Infrared spectra are collected as follows: light of discrete wavelengths from a laser is directed onto the tissue sample via glass fibers. Light scattered from the samples is collected in fibers and launched into a spectrometer. The plot of signal intensity as a function of wavelength can be then used to develop chemometric models to discriminate lipid-rich deposits from non-atherosclerotic tissue, and from atherosclerotic tissue that is predominantly fibrotic and from blood elements. This technique is incorporated into a thin catheter with similar dimensions to an IVUS catheter, and the intracoronary dwell time for analysis is similar to the broad experience with established techniques with proven safety, such as IVUS.

ELIGIBILITY:
Inclusion Criteria:

* >=18yrs and undergoing elective or non-emergent PCI of a de novo native coronary artery lesion
* Treatment plan (at time of consent and at time of intervention) must be to perform an intervention on no more than 2 lesions, where one is the culprit lesion and the other lesion requires revascularization at the discretion of the treating physician.
* Target lesion should have "low-risk" characteristics(defined by angiography)
* Subject must be able to read, understand and sign an approved informed consent form and follow protocol
* Female subjects of child bearing potential must have a negative serum pregnancy test prior to enrollment

Exclusion Criteria:

* Evidence of Clinical instability in the 6 hours before the procedure, or at any time during the procedure (72 hours stable post-STEMI)
* Angiographically Unsuitable Coronary and/or Lesion Morphology in the culprit vessel.
* A contraindication to anticoagulation or increased risk of bleeding.
* Clinically significant abnormal laboratory findings
* Presence of a drug eluting stent in the artery for experimental study prior to NIR measurement, unless all struts are covered by endothelium as documented by IVUS
* Elective PCI on or through bypass grafts or LIMA grafts
* Allergy or intolerance to aspirin or clopidogrel
* Planned use of laser ablation, rotational ablation, brachytherapy, or atherectomy device
* Enrollment or participation in any other medication trial within the previous 30 days
* Current enrollment participation or enrolled in another clinical trial
* Any other factor that the investigator feels would put the patient at increased risk if participating in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-01; Primary Completion 2007-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Waxman, MD, Principal Investigator — Lahey Clinic, Burlington, MA, USA
Locations (6):
- United States (5):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - William Beaumont Hospital, Royal Oak, Michigan
  - Columbia University Medical Center, New York, New York
  - Duke Medical Center, Durham, North Carolina
- Montreal Heart Institute, Montreal, Quebec, Canada

REFERENCES:
- [Result] Waxman S, Dixon SR, L'Allier P, Moses JW, Petersen JL, Cutlip D, Tardif JC, Nesto RW, Muller JE, Hendricks MJ, Sum ST, Gardner CM, Goldstein JA, Stone GW, Krucoff MW. In vivo validation of a catheter-based near-infrared spectroscopy system for detection of lipid core coronary plaques: initial results of the SPECTACL study. JACC Cardiovasc Imaging. 2009 Jul;2(7):858-68. doi: 10.1016/j.jcmg.2009.05.001. PMID 19608137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from patients presenting to the cardiac catheterization laboratory for scheduled elective percutaneous coronary intervention. Subject's medical history and angiographic coronary anatomy were used to evaluate eligibility.
Groups:
- Intravascular Coronary Imaging: Subjects undergoing intravascular ultrasound and near infrared spectroscopy imaging
Period: Overall Study
Arm/Group | Intravascular Coronary Imaging
Started | 106 (Subjects that signed consent and were subject to research procedures.)
7 Day Phone Contact | 99
1 Year Phone Contact | 89
Completed | 89
Not Completed | 17
Not completed — Lost to Follow-up | 6
Not completed — Physician Decision | 9
Not completed — Death | 1
Not completed — IVUS could not be performed. | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intravascular Coronary Imaging
Number analyzed (Participants) | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 65
  >=65 years | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.67 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 86
Region of Enrollment [Number; unit: participants]
  United States | 79
  Canada | 27

OUTCOME MEASURES:

1. Primary Outcome: Spectral Similarity
Description: Average spectral similarity of the spectra in a complete scan per patient as compared to the autopsy spectral data set.Clinical data was considered similar to autopsy data if average spectral similarity in each scan was >=67%, on a continuous range of 0%(different) to 100%(identical) similarity.
Time Frame: Baseline
Population: 58 Subjects were excluded from endpoint analysis for No NIRS data(17), Inadequate data per protocol(11), and Data Accessible during comparison set generation(30).A similarity success was met if >80% of the NIRS data for a subject was similar to the autopsy NIRS set.
Measure: Mean (95% Confidence Interval); unit: percent similarity
Arm/Group | Intravascular Coronary Imaging
Number analyzed (Participants) | 48
percent similarity | 83 [70 to 93]

2. Secondary Outcome: Review of Lipid Core Plaque of Interest Near Infrared Signals Observed at Baseline in Patients With Stable Angina vs Acute Coronary Syndromes
Description: This is an exploratory examination to determine if an association exists between the presence or characteristics of lipid core plaques of interest signals and the clinical designation of acute or stable coronary artery disease in enrolled subjects. The study is not powered for statistical significance for this outcome.
Time Frame: Baseline
Reporting Status: Not Posted

3. Secondary Outcome: Identification of Distinct Near Infrared Spectral Characteristics Associated With Special Coronary Artery Features Identified by Angiography and/or Intravascular Ultrasound and Patient Characteristics
Time Frame: Baseline
Reporting Status: Not Posted

4. Secondary Outcome: Clinical Cardiac Events Definitely Attributable to the Study Device That Occur From Enrollment to 7 Days Post Enrollment
Description: Major adverse cardiac events (MACE: myocardial infarction, cardiac surgery, death, cerebral vascular accident, coronary revascularization) will be evaluated for being categorized as Definitely attributable to the study device.
Time Frame: Baseline to 7 day
Population: All patients that were enrolled, intent to treat population, were evaluated for definite or probable relation to the investigational device. This includes 7 subjects that were not exposed to the investigational device.
Measure: Number; unit: participants
Arm/Group | Intravascular Coronary Imaging
Number analyzed (Participants) | 106
participants
  Myocardial Infarction | 0
  Target Vessel Revascularization | 0
  Death | 0
  Cerebral Vascular Accident | 0

5. Secondary Outcome: Cardiac Events That Occur Within 1 Year Post Enrollment Will be Examined for Link to Lipid Signals.
Description: Major adverse cardiac events (MACE: myocardial infarction, cardiac surgery, death, cerebral vascular accident, coronary revascularization) will be evaluated relation to baseline presence of lipid signals by near infrared spectroscopy. This study is not powered to reach statistical significance for this outcome.
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intravascular Coronary Imaging
Serious Adverse Events (participants affected / at risk) | 10
Other Adverse Events (participants affected / at risk) | 20
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Intravascular Coronary Imaging
Myocardial Infarction (Cardiac disorders) | 8/106 (9)
Cerebral Vascular Accident (Nervous system disorders) | 1/106 (1)
Death (Cardiac disorders) | 1/106 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Intravascular Coronary Imaging
Chest Pain/Shortness of Breath (Cardiac disorders) | 20/106 (28)

LIMITATIONS AND CAVEATS:
Technical limits of the prototype device factored into the data set reduction(28 patients).Data made available to evaluate handling of the device(30 patients) could not be prospectively evaluated for the primary endpoint of Spectral Similarity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days